CLINICAL TRIAL: NCT01700660
Title: Reperfusion-induced Self-antigen Excretion Following Major Liver Surgery
Acronym: RISE
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Megan J. Reiniers, PhD student at the Department of Surgery, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2012_238; NL41737.018.12 (Other: Central Committee on Research involving Human Subjects, the Netherlands)
Record Dates: First submitted 2012-10-03; First posted 2012-10-04 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Warm Hepatic Ischemia-reperfusion Injury

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 2 liver biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VIO: Patients operated under VIO.
- Control: Patients operated without VIO.

SUMMARY:
Major liver surgery often requires the surgeon to temporarily halt the afferent blood flow in order to prevent excessive blood loss. However, this predisposes the liver to a detrimental inflammatory response once the circulation is restored. Altogether, the effects that result from this temporary withdrawal of blood are known as ischemia and reperfusion (I/R) injury, and the extent to which this occurs determines the functional outcome of the liver after surgery.

Recently, it has become clear that (over)activation of the immune system forms the mainstay of I/R injury in the liver. More importantly, it has been shown in animal models that self-antigens, which are normal cellular constituents that become immunogenic mediators following their release from dying cells, are involved in the earliest stages of I/R injury of the liver. Clinical data on the release self-antigens in I/R injury are however scarce to date. Therefore, the aim of this study is to investigate the release of self-antigens in patients that undergo a major liver resection with or without withdrawal of the liver's blood flow. Also, the results will be correlated to genes involved in the inflammatory response as well as clinical parameters for liver damage and function.

DETAILED DESCRIPTION:
Rationale

Major liver surgery often requires the surgeon to temporarily halt the afferent blood flow in order to prevent excessive blood loss. Vascular inflow occlusion (VIO) however predisposes the liver to a detrimental inflammatory response once the circulation is restored. Altogether, the ramifications that result from this temporary withdrawal of oxygen supply are known as ischemia and reperfusion (I/R) injury, and the extent to which this occurs determines the functional outcome of the liver after surgery. Recently, it has become clear that (over)activation of the immune system forms the mainstay of hepatic I/R injury. More importantly, it has been shown in animal models that endogenous self-antigens, known as damage-associated molecular patterns (DAMPs), are released from stressed liver cells in the earliest stages of reperfusion and, as such, form the most proximal triggers of hepatic I/R injury. Clinical data on DAMP release following hepatic I/R are however scarce to date. Therefore, the aim of this study is to investigate DAMP release in patients that undergo a major liver resection with or without VIO and to correlate the results to the expression of acute- phase inflammatory response genes and routine clinical parameters for hepatocellular damage.

Objective

To investigate the release of damage-associated molecular patterns (DAMPs) following major hepatic resection with or without VIO and to correlate the outcomes to the acute inflammatory response and clinical parameters for hepatocellular damage.

Study design

The study is designed as an observational study. Because the decision to apply VIO is often made during surgery, patients will be allocated to a group postoperatively. Therefore, the inclusion of subjects in this study will continue until the calculated sample size of 15 patients has been reached in each group.

Study population

Eligible patients for participation in this study are those diagnosed with a malignant or benign hepatic tumor that are scheduled to undergo major hepatectomy (resection of ≥3 segments).

Main study parameters/endpoints

The primary endpoint of this study is defined as the effect of I/R on the release of DAMPs, measured in the systemic circulation. Secondary parameters constitute the expression of acute inflammatory response genes, AST, ALT, total bilirubin, and INR.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo a major liver resection for a benign or malignant hepatic tumor
* Signed informed consent obtained prior to any study-specific procedure
* ASA classification I-III

Exclusion Criteria:

* VIO <20 min
* ASA classification IV/V
* Emergency operations
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a malignant or benign hepatic tumor that are scheduled for a liver resection.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
DAMPs in systemic circulation | 8 hours
  Plasma DAMP levels will be determined perioperatively.

SECONDARY OUTCOMES:
Up regulation of acute inflammatory response genes | 1 hour
  Up regulation of acute inflammatory response genes will be determined in liver biopsy tissue (acquired intraoperatively) by means of qPCR.
Parenchymal damage | 8 hours
  Measured as plasma ALT and AST.
Liver function | 8 hours
  Assessed by means of total bilirubin levels and prothrombin time.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M. van Gulik, MD, PhD, Study Director — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Megan J. Reiniers, MSc, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Golen RF, van Gulik TM, Heger M. The sterile immune response during hepatic ischemia/reperfusion. Cytokine Growth Factor Rev. 2012 Jun;23(3):69-84. doi: 10.1016/j.cytogfr.2012.04.006. Epub 2012 May 17. PMID 22609105